CLINICAL TRIAL: NCT07386210
Title: Antihypertensive Effects of Rosmarinus Officinalis L. Infusion Supplements in Male Patients With Mild Hypertension : A Randomized Double-Blind Placebo-Controlled Study
Brief Title: Antihypertensive Effects of Rosmarinus Officinalis L. Infusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: awatef Sassi (Other)
Responsible Party: Sponsor-Investigator, awatef Sassi, PHD Assistant Professor at the Private Higher Institute of Nursing Sciences, Faculty of Medicine, Sousse
Organization: Faculty of Medicine, Sousse (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ROhypertension
Record Dates: First submitted 2026-01-11; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Hypertension Arterial
Keywords: Rosmarinus officinalis L; male hypertensive patients; hypertension; infusion
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bras 1 rosemary infusion (Experimental): Infusion prepared from 2g of rosemary leaves. Administered orally, 1 cup (100 mL) per day.
  Duration: 6 weeks.
  Interventions: Dietary Supplement: Rosemary extract infusion
- bras 2: placebo (Placebo Comparator): Infusion with color and taste similar to rosemary, without active extract
  Administered orally, 1 cup (100 mL) per day
  Duration: 6 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Rosemary extract infusion — Infusion prepared from 2g of rosemary leaves
  Administered orally, 1 cup (100 mL) per day
  Duration: 6 weeks
  Arms: Bras 1 rosemary infusion
Dietary Supplement: Placebo — Infusion with color and taste similar to rosemary, without active extract Administered orally, 1 cup (100 mL) per day Duration: 6 weeks
  Arms: bras 2: placebo

SUMMARY:
This study assessed the antihypertensive effect of rosemary tea through a placebo-controlled clinical study, angiotensin-converting enzyme (ACE) inhibition analysis, and in silico evaluation of interactions between rosemary bioactive compounds and the AT1R (Angiotensin II Type 1 Receptor).

A randomized, double-blind, placebo-controlled trial was conducted in 54 male patients with mild hypertension. Participants were assigned to receive either rosemary infusion (n = 27) or placebo (n = 23) for 45 days. Ambulatory blood pressure monitoring wass used to evaluate blood pressure parameters. Serum ACE activity was measured at baseline and after the intervention using FAPGG hydrolysis. Molecular docking simulations were performed using the Dock 4.2 software.

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged 28-65 years
* Mild hypertension, defined as systolic blood pressure (SBP) 140-159 mmHg and/or diastolic blood pressure (DBP) 90-99 mmHg, according to ESC/ESH 2018 guidelines
* No history of chronic diseases
* Not currently taking antihypertensive medications, other drugs, or dietary supplements
* Body mass index (BMI) within the screening range at recruitment
* Provided written informed consent

Exclusion Criteria:

* Secondary hypertension
* History of cardiovascular disease, diabetes mellitus, renal failure, autoimmune disease, or major gastrointestinal disorders
* Current use of medications affecting blood pressure
* Extreme body mass index (BMI) values
* Significant dietary changes or irregular physical activity in the previous six months
* Alcohol consumption or use of illicit drugs
* Inability or unwillingness to maintain usual diet and lifestyle during the study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — men with mild hypertension
Enrollment: 54 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Measurement of ambulatory blood pressure | 6 weeks
  ABPM was utilized to improve the accuracy of the clinical trial while minimizing the required number of participants. Blood pressure mea- surements were taken at the brachial artery using a Holter SunTech Medical Oscar 2 device (INC S07Air Port Blvd, Suite 117, Morrisville, NC, USA) to monitor BP over a 24-hour period. The device was set to record BP every 30 min during the day and every hour at night. The cuff was placed on the non-dominant arm, enabling the participants to carry on with their normal activities. They were instructed to stay still during cuff inflation.
  The sleep and wake times for programming the Holter device were established based on a question asked to the subjects during their visit. These measurements were recorded on Day 0 (D0) and Day 45 (D45) to assess the impact of the rosemary infusion on blood pressure. We assessed the following blood pressure parameters: 24-h, daytime, and nighttime SBP and DBP, mean blood pressure (MBP), heart rate (HR), and nocturnal d

SECONDARY OUTCOMES:
Determination of serm angiotensin-converting enzyme activity | 6 weeks
  Serum angiotensin-converting enzyme (ACE) activity was determined in men with grade 1 hypertension using serum samples collected at baseline and after six weeks of daily consumption of either rosemary infusions or a placebo. It was measured using the ACE Liquid reagent kit (Sentinel Diagnostics, Italy) on an automated clinical chemistry analyzer (Beckman Coulter AU 700, USA). The method is based on the enzymatic hydrolysis of the synthetic substrate FAPGG (furylacryloyl-phenylalanyl-glycyl-glycine). ACE catalyzes the cleavage of FAPGG, resulting in a decrease in absorbance at 340 nm, which is directly proportional to the ACE activity in the sample. Intra- and inter-assay precision coefficient of variation (CV) of the Beckman Coulter AU 700 Sentinel Diagnostics ACE values are 2.6% and 2.9%, respectively at 40 UI/L. The ACE activity measurement exhibits excellent linearity across the range of 5.8 U/L to 120 U/L, ensuring accurate quantification within this interval. Adults' normal ACE
Biochemical Analysis and Assessment | 6 weeks
  Blood samples were collected from the cubital vein of subjects both at baseline and after the study, following a 12-h fasting period. The samples were drawn into three distinct tubes: an EDTA-coated tube, a heparin-coated tube, and a sodium fluoride/potassium oxalate-coated tube. These samples were immediately subjected to centrifugation for 20 min at 3000 rpm, then stored at -80 ◦C until further analysis.
  Plasma aliquots were transferred to the biochemistry laboratory for the determination of various biochemical parameters and ionic con- stituents in the blood, including ASAT, ALAT, total bilirubin, direct bilirubin, γ-GT, alkaline phosphatase, cholesterol, triglycerides, HDL, LDL, glucose, urea, creatinine, uric acid, albumin, Na+, and K+. Ana- lyses were conducted at the Biochemistry Department of Farhat Hached Hospital in Sousse using the Unicell DXC 600 Synchron analyzer by Beckman Coulter. LDL cholesterol levels were calculated using the Friedewald formula.
Evaluation Perceived Benefits of Rosemary infusion | 6 weeks
  During the intervention period, participants were instructed to report any noticeable changes in health status associated with the use of rosemary infusion. This approach enabled the investigator to monitor safety and collect subjective observations related to the intervention.

OTHER OUTCOMES:
Binding affinity of rosemary phenolic compounds to hypertension target proteins assessed by molecular docking | 15 days
  Molecular docking simulations were carried out by the Auto Dock 4.2 program package (Trott and Olson, 2010). The 'XFEL structure of human Angiotensin Receptor' was sourced from Protein Data Bank (PDB code: 4YAY). The steps were done : add the missing hydrogens in addition to assigning the partial charges (Gasteiger). The AutoDock Tools were used to prepare the ligands and protein files (PDBQT). The optimization of all the geometries of ligands was conducted by using ACD (3D viewer) software (http://www.filefacts.com/acd3d-viewer-freeware-info) and the visualization and analysis of interactions were carried out via Discovery Studio 2017R2 (https://www.3dsbiovia. com/products/collaborative-science/biovia-discovery-studio/) and PyMOL 0.99rc6

CONTACTS AND LOCATIONS:
Locations (2):
- Tunisia (2):
  - Faculty of Medicine of Sousse, Sousse
  - Sassi, Sousse

IPD SHARING:
Plan to Share IPD: No